CLINICAL TRIAL: NCT00330343
Title: The Optimal Dose of Prophylactic Naloxone in Ameliorating Opioid Induced Side Effects in Children and Adolescents Receiving Intravenous Patient Controlled Analgesia (IVPCA) Morphine for Moderate to Severe Pain: A Pharmacodynamic, Pharmacokinetic, and Pharmacogenetic Study
Brief Title: Optimal Dose of Prophylactic Naloxone in Reducing Opioid-Induced Side Effects in Children/Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-03-31-02
Record Dates: First submitted 2006-05-24; First posted 2006-05-26 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Pain; Nausea; Pruritus
Keywords: morphine; naloxone; pediatrics; adverse effects; pain
MeSH Terms: conditions — Pain; Nausea; Pruritus | interventions — Naloxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Naloxone (Experimental): continuous infusion of naloxone administered in escalating dosing from 0.05 mcg/kg/hr to 1.65 mcg/kg/hour
  Interventions: Drug: naloxone

INTERVENTIONS:
Drug: naloxone — continuous infusion of naloxone administered in escalating dosing from 0.05 mcg/kg/hr to 1.65 mcg/kg/hour

SUMMARY:
This is an investigator initiated dose finding study designed to determine the optimal dose of naloxone to prevent or minimize the most common side effects induced by opioids, namely itching, nausea, and vomiting. Male and female inpatients of the Children's Center of the Johns Hopkins Hospital, who are greater than 6 and less than 18 years of age with acute, moderate to severe pain, and who are to be treated with intravenous Patient controlled analgesia (IVPCA) morphine will be eligible for inclusion in this study. Patients will be recruited by a study investigator prior to the initiation of IVPCA therapy. The majority of patients will be post operative patients, and will start therapy and the investigational drug in the Post Anesthesia Care Unit or the Pediatric Intensive Care Unit. The investigators plan on studying between 10 and 99, male and female patients over a 2 year period.

DETAILED DESCRIPTION:
In patients of all ages, opioids are the cornerstone of management of moderate to severe pain. Regardless of method of administration, all opioids produce unwanted side effects, including pruritus, nausea and vomiting, constipation, urinary retention, cognitive impairment, tolerance, dependence, and (rarely) respiratory depression. Based on the results of a previously completed randomized controlled trial, children and adolescents with moderate to severe pain, are now routinely treated in the Children's Center of the Johns Hopkins Hospital with a low dose naloxone infusion (0.25 mcg/kg/HOUR) whenever morphine intravenous patient controlled analgesia (IVPCA) or parent/nurse controlled analgesia (IVPNCA) is initiated. Although the previous study showed a marked reduction in the incidence and severity of pruritus and nausea, approximately a third of the patients still experience these side effects. The primary purpose of this study is to reduce this failure rate by determining if there is an optimal dose of naloxone to prevent opioid induced side effects as determined by a dose finding classic up down dose escalation method. The second aim is to determine the pharmacokinetics of morphine and naloxone and their metabolites at each of the naloxone infusion rates attempted. The investigators will measure morphine, naloxone, and their metabolites using a liquid chromatographic-electrospray ionization-tandem mass spectrometric method (LC/MS/MS). The final aim is to determine the pharmacogenetics of responders and non-responders using DNA isolated from patient blood. To accomplish this the investigators will need a single blood collection from patients currently being treated with IVPCA morphine and low dose intravenous naloxone.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients greater than 6 and less than 18 years of age with acute, moderate to severe pain who are to start treatment with IVPCA morphine as inpatients of the Children's Center of the Johns Hopkins Hospital

Exclusion Criteria:

* patients who require concomitant benzodiazepine administration
* allergic to opioids
* have been in an investigational drug trial within 1 month
* received opioids with in 7 days of the study
* parent with psychiatric illness which impairs their ability to provide consent parent who does not speak English

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2004-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron Yaster, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- John Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Maxwell LG, Kaufmann SC, Bitzer S, Jackson EV Jr, McGready J, Kost-Byerly S, Kozlowski L, Rothman SK, Yaster M. The effects of a small-dose naloxone infusion on opioid-induced side effects and analgesia in children and adolescents treated with intravenous patient-controlled analgesia: a double-blind, prospective, randomized, controlled study. Anesth Analg. 2005 Apr;100(4):953-958. doi: 10.1213/01.ANE.0000148618.17736.3C. PMID 15781505
- [Background] Gan TJ, Ginsberg B, Glass PS, Fortney J, Jhaveri R, Perno R. Opioid-sparing effects of a low-dose infusion of naloxone in patient-administered morphine sulfate. Anesthesiology. 1997 Nov;87(5):1075-81. doi: 10.1097/00000542-199711000-00011. PMID 9366459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 75 participants were consented, but only 64 participants participated in this study and were placed in the experimental arm.
Period: Overall Study
Arm/Group | Naloxone
Started | 64
Completed | 59
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Naloxone Side Effects
Description: incidence of nausea, vomiting, pruritus following naloxone infusion
Time Frame: 0-48 hours after infusion begins
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Naloxone
Number analyzed (Participants) | 64
participants | 32 [10 to 60]

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 32/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=59)
Nausea, Vomiting or pruritis (Gastrointestinal disorders) | 32 (59) — Nausea, vomiting, or pruritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No